CLINICAL TRIAL: NCT00639626
Title: Use of Levemir® Improves Metabolic and Clinical Status in CFRD
Brief Title: Use of Levemir® Improves Metabolic and Clinical Status in Cystic Fibrosis-related Diabetes (CFRD)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB07-00218
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Results first posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis Related Diabetes
MeSH Terms: interventions — Insulin Detemir; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levemir (Experimental)
  Interventions: Drug: insulin detemir [rDNA origin] injection

INTERVENTIONS:
Drug: insulin detemir [rDNA origin] injection — Starting dose of 0.1-0.3 units/kg/day in a once daily subcutaneous injection.
  Other Names: Levemir

SUMMARY:
This is a study to find out if Levemir® (a long acting or basal insulin) is safe and effective in treating cystic fibrosis related diabetes (CFRD).

DETAILED DESCRIPTION:
Cystic fibrosis (CF) related diabetes (CFRD) and glucose intolerance affects more than 50%-75% of teens and adults with CF. The 1998 North American CF Foundation on CFRD categorized the disease differently than other types of diabetes: CFRD with fasting hyperglycemia (FH), CFRD without FH and transient CFRD. The outcome of this consensus conference was the use of insulin as the only recommended treatment of CFRD. Although the conference report mandated treatment for CFRD with FH, treatment was not mandated for the other types of CFRD, the choice to treat was left to the clinician's discretion. However, insulin was the only recommended therapy for all types of CFRD. Although some clinicians have used basal bolus regimens as the insulin management, many still use NPH. Given the need for CF patients to eat many frequent meals and snacks to maintain their weight, use of NPH insulin rarely renders good glycemic control. A basal bolus regimen is much more physiologic and would allow good glycemic control even with frequent meals and snacks. To date, there are no studies documenting safety and efficacy of true basal insulin, or a basal bolus regimen. Furthermore, protein catabolism and excessive muscle loss has been well documented in CF patients, both in those with and those without, glucose intolerance. Studies by our group and others have documented that a major reason for the catabolism is resistance to insulin's anti-catabolic effects on protein turnover. Thus, there is potential clinical benefit of improving muscle mass and general health by insulin treatment even for CF patients who do not have fasting hyperglycemia. A non-peaking basal insulin would be the only reasonable choice, yet studies are lacking. Our overall goal is to study the safety and efficacy of LevemirTM for the improvement of glycemic control of patients with CFRD. As a second goal, we will explore the ability of this basal insulin to improve protein catabolism and muscle mass. The study will be conducted as a six month trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CFRD by oral glucose tolerance test (OGTT) who are medically stable. Medical stability will be defined as:

  * No hospital admission for six weeks or more before the study
  * No oral or intravenous antibiotics for at least six weeks preceding the study (subjects will be allowed to use low doses of inhaled corticosteroids).

Exclusion Criteria:

* Use of oral or intravenous corticosteroid medications within six weeks of the study.
* Evidence of clinically significant liver disease.
* Colonization with Burkholderia cepacia.
* Colonization with Aspergillus.
* Pregnancy.
* Medically unstable (stability defined above).

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana S. Hardin, MD, Principal Investigator — OSU, Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Hardin DS, Moran A. Diabetes mellitus in cystic fibrosis. Endocrinol Metab Clin North Am. 1999 Dec;28(4):787-800, ix. doi: 10.1016/s0889-8529(05)70102-x. PMID 10609120
- [Background] Hardin DS, LeBlanc A, Para L, Seilheimer DK. Hepatic insulin resistance and defects in substrate utilization in cystic fibrosis. Diabetes. 1999 May;48(5):1082-7. doi: 10.2337/diabetes.48.5.1082. PMID 10331413
- [Background] Moran A, Milla C, Ducret R, Nair KS. Protein metabolism in clinically stable adult cystic fibrosis patients with abnormal glucose tolerance. Diabetes. 2001 Jun;50(6):1336-43. doi: 10.2337/diabetes.50.6.1336. PMID 11375334
- [Background] Moran A, Doherty L, Wang X, Thomas W. Abnormal glucose metabolism in cystic fibrosis. J Pediatr. 1998 Jul;133(1):10-17. doi: 10.1016/s0022-3476(98)70171-4. No abstract available. PMID 9672504
- [Background] Cucinotta D, Arrigo T, De Luca F, Di Benedetto A, Lombardo F, Scoglio R, Sferlazzas C, Magazzu G. Metabolic and clinical events preceding diabetes mellitus onset in cystic fibrosis. Eur J Endocrinol. 1996 Jun;134(6):731-6. doi: 10.1530/eje.0.1340731. PMID 8766944
- [Background] Nir M, Lanng S, Johansen HK, Koch C. Long-term survival and nutritional data in patients with cystic fibrosis treated in a Danish centre. Thorax. 1996 Oct;51(10):1023-7. doi: 10.1136/thx.51.10.1023. PMID 8977604

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PI left institution suddenly in 2010 and studies were closed. Study records for participants cannot be located and possibly have been destroyed.
Period: Overall Study
Arm/Group | Levemir
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: PI left institution suddenly in 2010 and studies were closed. Study records for participants cannot be located and possibly have been destroyed.
Arm/Group | Levemir
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Blood Sugar
Time Frame: 6 months
Population: as for baseline characteristics
Arm/Group | Levemir
Number analyzed (Participants) | 0

2. Secondary Outcome: Lean Body Mass
Time Frame: 6 months
Population: as for baseline characteristics
Arm/Group | Levemir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: PI left institution suddenly in 2010 and studies were closed. Study records for participants cannot be located and possibly have been destroyed.
Arm/Group | Levemir
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes